CLINICAL TRIAL: NCT05745090
Title: Performance of NT-proBNP in Risk Stratification for Cardiovascular Events and Mortality in Patients With Diabetes (PISCES)
Brief Title: N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) in Type 2 Diabetes Mellitus
Acronym: PISCES
Status: Active, not recruiting | Type: Observational
Sponsor: Singapore General Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PISCES2022
Record Dates: First submitted 2023-02-09; First posted 2023-02-27 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Type2diabetes; Heart Failure; Cardiovascular Complication
Keywords: Diabetes; Risk prediction
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1.5 - 2.0 ml of serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
More than 400 million people have type 2 diabetes (T2D) globally, and the burden of diabetes-related cardiovascular complications is increasing. Cardiovascular disease (CVD) affects approximately one-third of all individuals with T2D and accounts for half of all deaths in this population despite major advances in the treatment of the disease. Among the different types of CVD, heart failure (HF) is frequently the first CVD manifestation in individuals with T2D. Although the link between T2D and CVD is widely recognised, the absolute risk of cardiovascular events varies among individuals with T2D. As such, effective risk-stratification tool that accurately identify T2D patients at the highest risk of developing incident or recurrent cardiovascular (CV) events is needed.

B-type natriuretic peptide (BNP) and its inactive N-terminal precursor NT-proBNP are biomarkers of myocardial stress. They been shown to incrementally improve predictive discrimination of death and CV events in high-risk individuals with T2D.

An NT-proBNP-based CVD/HF risk stratification strategy has not been prospectively tested in the multi-ethnic T2D population in Singapore. In this study, we aim to:

1. Evaluate the predictive value of NT-proBNP for death and CV events compared to traditional risk markers [e.g. HbA1c, albuminuria, high sensitivity C-reactive protein (hsCRP), high sensitivity troponin-T (hsTnT)] in a cohort of T2D patients with or without established CVD (defined as ischaemic heart disease, myocardial infarct, unstable angina, prior coronary artery revascularisation, stroke, transient ischaemic attack or PAD) attending a tertiary diabetes care centre. (Patients with history of HF will be excluded.)
2. Compare the performance of NT-proBNP as a single biomarker for CV risk prediction to risk scoring algorithms in T2D patients.

DETAILED DESCRIPTION:
This is a prospective single-site, observational study to evaluate the predictive value of NT-proBNP for death and CV events compared to traditional CV risk markers (e.g., HbA1c, albuminuria, hsCRP and hsTnT) in T2D patients with or without established CVD (defined as ischaemic heart disease, myocardial infarct, unstable angina, prior coronary artery revascularisation, stroke, transient ischaemic attack or PAD). Patients with history of HF will be excluded. The study will also compare the performance of NT-proBNP as a single biomarker for CV risk prediction to other risk scoring algorithms such as UK Prospective Diabetes Study (UKPDS) risk engine, Risk Equations for Complications Of Type 2 Diabetes (RECODe) and University of Hong Kong-Singapore (HKU-SG) risk scores.

The study will prospectively recruit 1200 adults (aged 40 and above) with T2D from Singapore General Hospital (SGH) over a period of 18 months. Informed consent will be obtained from patients before the start of any procedures. There will be 1 baseline visit to collect demographic information, and clinical and laboratory data. Baseline point-of-care echocardiography will also be performed for all patients. All patients will subsequently be observed over 5 years for the occurrence of death or CV events through monitoring of electronic health records (EHR) and telephone contacts.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes (T2D) of at least 6 months' duration
2. Age 40 and older

Exclusion Criteria:

1. Known history of heart failure (self-reported and medical records review)
2. Estimated glomerular filtration rate (eGFR) <15 ml/min/1.73m2 [using the CKD-Epidemiology Collaboration (CKD-EPI) 2021 equation for glomerular filtration rate] based on the last known eGFR within 12 months of study recruitment)
3. Renal replacement therapy
4. Systemic treatment with corticosteroids or immunosuppressants
5. Pregnant or nursing women
6. Active cancer disease
7. Serious disease with life expectancy <1 year as judged by the doctor
8. Any condition that, in the investigator's opinion, would interfere with a subject's ability to comply with study protocol or procedures

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes mellitus age 40 and above, without known history of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with composite endpoint based on first occurrence of all-cause death or cardiovascular events | 5 years
  Composite endpoint based on the first occurrence of all-cause death or CV events consisting of a composite of non-fatal myocardial infarction, non-fatal stroke, unplanned hospitalisation for heart failure (HHF), coronary revascularisation (PCI or CABG), non-traumatic lower limb amputation, or lower limb arterial revascularisation (surgical or endovascular).

SECONDARY OUTCOMES:
Number of participants with cardiovascular (CV) death | 5 years
  Cardiovascular death consists of death due to acute myocardial infarction, sudden cardiac death, death due to heart failure, stroke, CV procedure, CV hemorrhage or other CV cause.
Number of participants with all-cause death | 5 years
  Death due to any cause.
Number of unplanned hospitalization for heart failure (HHF) | 5 years
  Refers to heart failure event that was a cause of hospitalization (primary or contributing) following baseline visit.
Number of participants with 4-point major adverse cardiovascular event (MACE) | 5 years
  Include CV death, non-fatal myocardial infarction, non-fatal stroke, unplanned HHF
Number of participants with all-cause hospitalization | 5 years
  Include emergency, unplanned or non-elective all-cause hospitalizations

OTHER OUTCOMES:
Proportion of study subjects with reduced left ventricular systolic function | Baseline
  Proportion of study subjects with reduced left ventricular systolic function
Proportion of study subjects with reduced left ventricular diastolic function | Baseline
  Proportion of study subjects with reduced left ventricular diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Yong Mong Bee, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Background] Matheus AS, Tannus LR, Cobas RA, Palma CC, Negrato CA, Gomes MB. Impact of diabetes on cardiovascular disease: an update. Int J Hypertens. 2013;2013:653789. doi: 10.1155/2013/653789. Epub 2013 Mar 4. PMID 23533715
- [Background] Birkeland KI, Bodegard J, Eriksson JW, Norhammar A, Haller H, Linssen GCM, Banerjee A, Thuresson M, Okami S, Garal-Pantaler E, Overbeek J, Mamza JB, Zhang R, Yajima T, Komuro I, Kadowaki T. Heart failure and chronic kidney disease manifestation and mortality risk associations in type 2 diabetes: A large multinational cohort study. Diabetes Obes Metab. 2020 Sep;22(9):1607-1618. doi: 10.1111/dom.14074. Epub 2020 Jun 3. PMID 32363737
- [Background] Hobbs FD, Jukema JW, Da Silva PM, McCormack T, Catapano AL. Barriers to cardiovascular disease risk scoring and primary prevention in Europe. QJM. 2010 Oct;103(10):727-39. doi: 10.1093/qjmed/hcq122. Epub 2010 Aug 4. PMID 20685842
- [Background] Malachias MVB, Jhund PS, Claggett BL, Wijkman MO, Bentley-Lewis R, Chaturvedi N, Desai AS, Haffner SM, Parving HH, Prescott MF, Solomon SD, De Zeeuw D, McMurray JJV, Pfeffer MA. NT-proBNP by Itself Predicts Death and Cardiovascular Events in High-Risk Patients With Type 2 Diabetes Mellitus. J Am Heart Assoc. 2020 Oct 20;9(19):e017462. doi: 10.1161/JAHA.120.017462. Epub 2020 Sep 23. PMID 32964800